CLINICAL TRIAL: NCT05995574
Title: Improving Clinician Communication About Contraception Using Teen and Parent Avatars
Brief Title: Avatar Contraception Communication Training
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Jenny Francis, Associate Professor, University of Texas Southwestern Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: Pending funding
Record Dates: First submitted 2023-05-16; First posted 2023-08-16 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Communication
Keywords: Adolescent; Contraception; Training
MeSH Terms: conditions — Communication

STUDY DESIGN:
Intervention Model Description: single intervention arm with pre- and post- evaluation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Avatar training (Experimental): One hundred physician learners will train with the avatar communication training tool as a behavioral intervention. Before the training (T0), the learners will complete a pre-survey to assess their baseline confidence. At the start of training, after a brief introduction and orientation to the tool, the learners will complete a 10-min uninterrupted scenario with a teen-parent avatar dyad about a contraception scenario. After the initial scenario (T1), the learner will pause and complete an assessment to evaluate use of SDM (Shared decision making) skills and PCCC (person-centered contraceptive counseling). Then, the learner will train for an hour with the tool. At the end (T2), the learner will complete another uninterrupted scenario and evaluate their confidence, SDM, and PCCC skills.
  Interventions: Behavioral: avatar communication training

INTERVENTIONS:
Behavioral: avatar communication training — Avatar simulates a mother and a daughter for the pediatrician to practice communication about contraception.

SUMMARY:
In order to support the desire of most adolescents to delay pregnancy (parenting) until their own adulthood, pediatricians must be comfortable and skilled in having reproductive health conversations with adolescents and the mothers of adolescents. Advocates for Youth (AFY), a national, youth-facing, well-established, non-profit, is known for innovative sexual and reproductive health programs. AFY successfully implemented a virtual simulation for schoolteachers to practice sex education scenarios by interacting with culturally diverse student avatars. We will partner with AFY to adapt their novel simulation-based approach to train medical residents in using SDM with youth and parent avatars. Our long-term goal is to build clinician confidence in SDM and actual skills via simulation training with dyadic avatars. We will also explore how evaluation of clinician communication skills varies from youth-, parent-, and clinician-viewpoints.

DETAILED DESCRIPTION:
Specific Aims seek to (1) iteratively adapt and refine the simulation training (1a) and measurement tools (1b) with three community advisory boards (CAB) of separate groups of teens, parents, and clinicians; and (2) conduct a proof-of-concept pre-post evaluation of clinician confidence in counseling dyads after one-time exposure to the simulation (n=100 medical residents). We will record residents' communications in the simulation and a subset of clinicians, parents, and adolescents from each CAB will evaluate residents' SDM skills via the Person-Centered Contraception Counseling (PCCC) scale. Hypothesis: Most medical residents (75%) will self-report improvement or stability in confidence with high acceptability of the simulation training. We will explore 1) overall concordance between self- and expert-reported evaluation outcomes (SDM skills, PCCC scale); 2) compare the distribution of each evaluation item by evaluator; and 3) explore correlations between scales by evaluator. Impact: This proof-of-concept study, co-developed and co-evaluated with community members and families, fills a gap in communication training to inform a future fully powered ORBIT stage 3 efficacy trial to test actual triadic communication in the real-world with comparator groups of medical residents across national training programs.

ELIGIBILITY:
Inclusion Criteria (providers):

* Providers (medical residents, fellows, attendings)
* Recruited from the Adolescent and Young Adult (AYA) Medicine Clinic at Children's Medical Center of Dallas.

Exclusion Criteria:

* Unable to speak or read in Spanish/English

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 166 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2030-06-30 (Estimated); Study Completion 2030-06-30 (Estimated)

PRIMARY OUTCOMES:
Questionnaire | Change from baseline (T0) at 0 hours, and end of training (T2) at 2 hours
  Multiple questions will be aggregated to arrive at one reported value to determine "improvement or stability in confidence" in shared decision-making communication.

SECONDARY OUTCOMES:
Acceptability Questionnaire | At end of study (T2) at 2-hours
  Weiners implementation outcome measure Acceptability of Intervention Measure (AIM). Items are measured on a 5-point Likert scale (Completely Disagree-Completely Agree). Score is calculated mean with the higher score meaning acceptability.
Questionnaire | Change from start (T1) at 20 minute to end of training (T2) at 2 hours
  Self-reported evaluation of a behavioral outcome (SDM (shared decision-making) skills and PCCC (person-centered contraception counseling) from start (T1) to end of training (T2)
Questionnaire | Change from start (T1) at 20 minute to end of training (T2) at 2 hours
  Expert evaluation of behavioral outcome (SDM (shared decision-making) skills and PCCC (person-centered contraception counseling) from start (T1) to end of training (T2)

CONTACTS AND LOCATIONS:
Overall Officials: Jenny KR Francis, MD, Principal Investigator — UTSouthwestern
Locations (2):
- United States (2):
  - Childrens Health Adolescent and Young Adult Medicine (AYA) Clinic, Dallas, Texas
  - UT Southwestern Medical Center, Dallas, Texas

IPD SHARING:
Plan to Share IPD: Yes
This study will collect 100 pre-post-surveys from clinicians in training, and 300 survey evaluations of video recordings. The study protocol, data tracking forms, survey, code book, data dictionary and a glossary of domain-specific terms will be shared in a portable document format (PDF).
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: 12mo after collection and available per Institutional Review Board standards
Access Criteria: All deidentified study data that are not designated as restricted use will be made available as public use data to the research community via DSDR.